CLINICAL TRIAL: NCT02761304
Title: Assessment of the Interests of Mesure of Ultrasound Engagement on the Cesarean Rate :Study Eng - Echo Randomized Comparative Prospective Study Multicenter Center Open
Brief Title: Assessment of the Interests of Mesure of Ultrasound " Angle of Progression " on the Cesarean Rate :a Randomized Comparative Prospective Study Multicenter Center Open
Acronym: eng - echo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2012-A01693-40; 2012-53 (Other: AP-HM)
Record Dates: First submitted 2016-05-02; First posted 2016-05-04 (Estimated); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Caesarean Rate
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- ultrasound results given to obstetrical practionnair (Experimental)
  Interventions: Procedure: Ultrasound
- ultrasound results shaded to obstetrical practionnair (Other)
  Interventions: Procedure: Ultrasound

INTERVENTIONS:
Procedure: Ultrasound

SUMMARY:
The reduction in the rate of caesarean section is a major public health issue, it has reached 21% in 2010 Fance. Indeed complications to expect during pregnancy and childbirth increase doubles the risk of fetal morbidity, néonatal and maternal history of when césareinne. recommendations for clinical practice (RPC) to "scarred uterus" are being drafted under the auspices of the National College of obstetrics and gynecology (CNGOF) well highlighting the health problem public this represents. During 2011, 15% of the 2,700 patients who have recently given birth to the north of Marseille Hospital were carriers of a scarred uterus (internal data).The objective of the obstetrician is to ensure the welfare mother and fetus at the end of pregnancy and childbirth. To do this, the realization of a work being cesarean allows in some cases to reduce neonatal morbidity related to workflow especially in case of abnormal fetal pericardial pace that suggest fetal hypoxia. However, a significant number of caesarean section is performed by the side of caution during the second part of the work to a suspicion of non-engagement of the fetal presentation. These caesareans are indicated, rightly, before a clinical doubt about the height of the engagement of the fetal presentation in order to avoid making a difficult instrumental delivery, potentially harmful to the mother (perineal tear 3rd and 4th degree) and fetus (head injury, intracranial hemorrhage, cephalohematoma). A prospective study published in the Lancet estimated 37% error percentage attributable to the clinical examination in case of doubt on the commitment of presenatation fœtale. The CNGOF held through PRC publication what to do in case of obstetric clinical doubt about the commitment of the fetal presentation and "not recommended" no show against an instrumental extraction in this situation (RPC 2008).

Ultrasound has revolutionized pregnancy monitoring. Its routine use has in other prenatal diagnosis of fetal pathologies, it is the other reference screening tool of the most common obstetric pathology, preterm labor. Its use became widespread in the delivery room, the presence of an ultrasound machine is recommended by the decrees of perinatal care in maternity hospitals performing more than 1,500 deliveries per year. It is natural for conducting ultrasound during labor has emerged, first to help identify the variety of the presentation of the fetal head and then more recently in aid to instrumental delivery. Several studies have shown that ultrasound had a sensitivity of commitment over 90% for predicting the success of instrumental extraction and a vaginal delivery.

To our knowledge, to date, there is no study that investigated the benefit of ultrasound commitment to reduce the rate of cesarean section during labor. To answer this question, we want to show that making a commitment in case of diagnostic ultrasound of doubt about the level of engagement of the fetal head (4% of births) reduces by 30% the rate of caesarean section fully dilated.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy normal evolution> 37 weeks gestation
* Patient in labor with ruptured membranes, cephalic presentation, full dilatation since 2H, with doubts on clinical examination on the level of engagement of the fetal head in the maternal pelvis (0, +1, +2)

Exclusion Criteria:

* Abnormal fetal heart rate or suspected fetal acidosis on a scale pH
* No maternal indication for vaginal delivery or instrumental delivery

  * History of perineal tearing the 4th degree
  * Crohn's disease with involvement of the anal sphincter
* No fetal indication for instrumental delivery (suspected fetal thrombocytopenia)
* Other than fetal cephalic presentations

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-06; Primary Completion 2015-09-09 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Caesarean rate | 2 years
  Demonstrate that achieving a so-called "engagement" ultrasound (mesurement of angle of progression) to reduce 30% cesarean rate in the second stage of labor in case of doubt about the level of commitment of fetal presentation. The primary endpoint is the rate of caesarean section.

SECONDARY OUTCOMES:
Numbers of haemorrhage | 2 years
perineal tears of 3 and 4th degree | 2 years
  perineal wounds

OTHER OUTCOMES:
Apgar scoring | 2 years
  Side effects with short term fetal complication

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — ASSISTANCE PUBLIQUE DE MARSEILLE
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haumonte JB, Blanc J, Castel P, Mace P, Auquier P, d'Ercole C, Bretelle F. Uncertain fetal head engagement: a prospective randomized controlled trial comparing digital exam with angle of progression. Am J Obstet Gynecol. 2022 Oct;227(4):625.e1-625.e8. doi: 10.1016/j.ajog.2022.04.018. Epub 2022 Apr 19. PMID 35452654